CLINICAL TRIAL: NCT01745081
Title: Comparison of the Efficacy Between 20% Mannitol and 3% Hypertonic Saline, Given as a Bolus at the Beginning of Elective Supratentorial Craniotomy for Tumor Resection, in Favoring Cerebral Relaxation Evaluated by a Sub-dural Intracranial Pressure Measurement.
Brief Title: Comparison of 20% Mannitol and 3% Hypertonic Saline for Cerebral Relaxation During Elective Supratentorial Craniotomies
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Stéphane Coutu, Principal study investigator, Centre de recherche du Centre hospitalier universitaire de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Study on cerebral relaxation
Record Dates: First submitted 2012-12-05; First posted 2012-12-07 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Osmotherapy; Intracranial Pressure
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol (Experimental): Bolus mannitol 20% at skin incision
  Interventions: Drug: 20% mannitol bolus administration
- Hypertonic saline (Experimental): Hypertonic saline 3% at skin incision
  Interventions: Drug: Hypertonic saline 3% bolus administration

INTERVENTIONS:
Drug: 20% mannitol bolus administration
  Arms: Mannitol
Drug: Hypertonic saline 3% bolus administration
  Arms: Hypertonic saline

SUMMARY:
Mannitol 20% has long been used to treat elevated intracranial hypertension in trauma and intensive care settings. More recent data indicate that hypertonic saline may be as effective or more effective than mannitol for this purpose, with possible fewer side effects.

This study compares both agents in favoring cerebral relaxation during elective supratentorial procedures for tumor resection.

Study hypothesis: 3% hypertonic saline will provide better cerebral relaxation with fewer side effects than 20% mannitol.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective supratentorial craniotomy for tumor resection
* Presumed preoperative diagnosis of : astrocytoma (any grade), meningioma (any sub-type) or cerebral metastasis (any primary neoplasm)

Exclusion Criteria:

* Age < 18 years
* Reintervention
* Glasgow coma scale < 13
* Emergency surgery or American Association of Anesthesiologists physical status class 4 or 5
* Prone or lateral positioning
* Hypo or hypernatremia (serum sodium below 135 or above 150 meq/L)
* Osmotherapy (either mannitol or hypertonic saline) given in the last 24 hours
* Congestive heart failure (LVEF < 40% or restrictive diastolic dysfunction on echocardiography)
* Chronic renal failure (creatinine clearance < 30 ml/min)
* Pregnancy
* Obesity (BMI > 40)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Sub-dural intracranial pressure | In average 30-60 minutes after intervention, just before dura mater opening
  Sub-dural measure of intracranial pressure to evaluate cerebral relaxation

SECONDARY OUTCOMES:
Subjective evaluation of cerebral relaxation | In average 30-60 minutes after intervention, just after dura mater opening
  Subjective evaluation by the surgeon of cerebral relaxation on a 4 point scale
Serum lactate | In average 5-8 hours after intervention, upon arrival in the intensive care unit
  Serum lactate measurement to assess tissue perfusion during the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada